CLINICAL TRIAL: NCT05834816
Title: Neural Mechanisms of Negative Affect and Neurofeedback in Anorexia Nervosa
Brief Title: Stress and Neurofeedback in Anorexia Nervosa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding received
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 805807
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral (Experimental): Negative Affect Task
  Interventions: Behavioral: Negative Affect Task

INTERVENTIONS:
Behavioral: Negative Affect Task — fMRI stress task
  Other Names: Functional Magnetic Resonance Brain Imaging Stress Task

SUMMARY:
Anorexia nervosa (AN) and atypical AN (AAN) are severe psychiatric illnesses associated with high disease burden including high treatment costs and excessive mortality rates. Primary characteristics of AN and AAN are food restriction, associated fear of weight gain, and a disturbance in how one's body weight or shape is experienced.The underlying neural mechanisms for the core illness behaviors of food restriction and body size overestimation in anorexia nervosa and atypical anorexia nervosa are not well understood.

This project will use neurofeedback and advanced psychophysical methods to assess and moderate the neural and behavioral responses to stress and relate those results to the naturalistic environment. The results will guide the development of novel interventions.

DETAILED DESCRIPTION:
The overall strategy is a cross-sectional study, involving 3 subject groups, each subject studied on two study days (one negative and one neutral affect day, randomized), one week apart; on both study days subjects will undergo functional magnetic resonance imaging (fMRI) during which they complete tasks for 1) neurofeedback-reward learning and 2) body size estimation. Before and after each scan, and in the week between scans, subjects will be assessed for positive and negative affect and how it affects food intake.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls (HC)

* Individuals aged 18-45 years
* Healthy body weight between 90 and 110 % average body weight since puberty.
* Regular monthly menstrual cycle (if applicable)
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* All ethnic backgrounds
* English is primary language spoken

Anorexia Nervosa (AN)

* Age 18-45 years old
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* All ethnic backgrounds
* Current diagnosis of anorexia nervosa, including being underweight, will have a severe fear of weight gain, body image distortion and absence of the menstrual cycle over three consecutive months.
* English is primary language spoken

Atypical Anorexia Nervosa (AAN)

* Age 18-45 years old
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* All ethnic backgrounds
* Meets the criteria for anorexia nervosa except despite significant weight loss, the individual's weight is within or above the normal range
* English is primary language spoken

Exclusion Criteria:

Healthy Controls (HC)

* Current pregnancy or breast feeding within last 3 months
* First degree relative with current or past eating disorder
* Psychiatric Medication use such as selective serotonin reuptake inhibitors (SSRIs), atypical antipsychotics, etc.
* Past or present Axis I psychiatric disorder including substance or alcohol use disorder as determined through structured clinical interview
* History of significant head trauma
* Indication of intellectual disability or autism spectrum disorder
* Major Medical illness that requires medication or have significant impact on subject's life such as: diabetes, Alzheimer's disease or dementia, stroke, learning disability, mobility disorders, cancer, high blood pressure, etc. (to be determined through biological screening form and interview with principal investigator (PI)
* Recent history of suspected substance abuse or a lifetime history of psychostimulant abuse and/or dependence
* Contraindications to magnetic resonance imaging (MRI) including metal implants or braces (as determined through fMRI screening form)

Anorexia Nervosa (AN)

* Pregnancy or breast feeding within last 3 months
* Lifetime history of bipolar I disorder or psychosis
* Current substance abuse or dependence in the past 3 months
* Psychotic illness/other organic brain syndromes, dementia, somatization disorders or conversion disorders
* Physical conditions (e.g., diabetes mellitus, pregnancy) known to influence eating or weight
* History of significant head trauma
* Indication of intellectual disability or autism spectrum disorder
* Electrolyte, blood count or kidney or liver function abnormalities
* Contraindications to MRI including metal implants or braces (as determined through fMRI screening form)

Atypical Anorexia Nervosa (AAN)

* Pregnancy or breast feeding within last 3 months
* Lifetime history of bipolar disorder or psychosis
* Current substance abuse or dependence in the past 3 months
* Psychotic illness/other organic brain syndromes, dementia, somatization disorders or conversion disorders
* Physical conditions (e.g., diabetes mellitus, pregnancy) known to influence eating or weight
* History of significant head trauma
* Indication of intellectual disability or autism spectrum disorder
* Electrolyte, blood count or kidney or liver function abnormalities
* Contraindications to MRI including metal implants or braces (as determined through fMRI screening form)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) brain activation in response to stress during a taste reward task | Difference in brain response between the neutral and stress condition, up to 9 days
  Activation in the brain during a taste reward task will be measured using functional MRI (fMRI) after a neutral and stressful task.
Functional Magnetic Resonance Imaging (fMRI) brain activation in response to stress during a body size estimation task | Difference in brain response between the neutral and stress condition, up to 9 days
  Activation in the brain during a body size estimation task will be measured using functional MRI (fMRI) after a neutral and stressful task.

SECONDARY OUTCOMES:
Ecological Momentary Assessment (EMA) | Up to 9 days
  Ecological Momentary Assessment (EMA) will be used to test food restriction and body size estimation in the natural environment and in relation to daily stress.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frank GKW, Shott ME, Stoddard J, Swindle S, Pryor TL. Association of Brain Reward Response With Body Mass Index and Ventral Striatal-Hypothalamic Circuitry Among Young Women With Eating Disorders. JAMA Psychiatry. 2021 Oct 1;78(10):1123-1133. doi: 10.1001/jamapsychiatry.2021.1580. PMID 34190963
- [Background] Gardner RM, Bokenkamp ED. The role of sensory and nonsensory factors in body size estimations of eating disorder subjects. J Clin Psychol. 1996 Jan;52(1):3-15. doi: 10.1002/(SICI)1097-4679(199601)52:13.0.CO;2-X. PMID 8682909
- [Background] Gardner RM, Boice R. A computer program for measuring body size distortion and body dissatisfaction. Behav Res Methods Instrum Comput. 2004 Feb;36(1):89-95. doi: 10.3758/bf03195553. PMID 15190703
- [Background] Misaki M, Phillips R, Zotev V, Wong CK, Wurfel BE, Krueger F, Feldner M, Bodurka J. Real-time fMRI amygdala neurofeedback positive emotional training normalized resting-state functional connectivity in combat veterans with and without PTSD: a connectome-wide investigation. Neuroimage Clin. 2018 Aug 19;20:543-555. doi: 10.1016/j.nicl.2018.08.025. eCollection 2018. PMID 30175041